CLINICAL TRIAL: NCT04872218
Title: A Double-blind Randomized Controlled Trial of 6-month of Abatacept vs Placebo as Adjuvant to Peanut Oral Immunotherapy to Induce Immunologic Changes in Patients With Severe Persistent Peanut Allergy
Brief Title: Adjuvant Treatment With Abatacept to Promote Remission During Peanut Oral Immunotherapy
Acronym: ATARI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Philippe Bégin (Other)
Responsible Party: Sponsor-Investigator, Philippe Bégin, Associate professor, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CITO-2021-01
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Peanut Allergy
Keywords: Peanut allergy; Abatacept; Oral immunotherapy
MeSH Terms: conditions — Peanut Hypersensitivity | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abatacept (Experimental)
  Interventions: Drug: Abatacept; Other: Peanut oral immunotherapy
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Other: Peanut oral immunotherapy

INTERVENTIONS:
Drug: Abatacept — 24 week treatment of IV abatacept following recommended dosages from the monograph
  Arms: Abatacept
Drug: Placebo — 24 week treatment of IV placebo following recommended dosages from the abatacept monograph
  Arms: Placebo
Other: Peanut oral immunotherapy — Peanut oral immunotherapy, following a patient-driven protocol, starting 24 to 72h after the first administration of abatacept or placebo.

SUMMARY:
This is a phase 2a, multi-center, randomized and double-blind placebo-controlled trial comparing 24 weeks of abatacept versus placebo used as adjuvant to oral immunotherapy to induce remission in adolescents and adults with persistent severe peanut allergy.

This is a proof-of-concept trial in which the primary outcome will be the suppression of the initial peanut specific IgE surge during OIT, which is used as a proxy outcome of peanut allergy remission.

Adolescents and adults with persistent severe peanut allergy (n=14) will be randomized to either abatacept or placebo at a ratio 1:1 for a total period of 24 weeks. Peanut oral immunotherapy will be initiated the day following the first administration of the investigational product. Sustained tolerance to peanut will be assessed at 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 14 to 50 years old at screening visit
* History of IgE mediated allergy to peanut protein
* ImmunoCAP IgE level > 50 kU/L for peanut;
* Total IgE level < 5000 kU/L
* Willing to comply to all study requirements during participation in the study;

Exclusion Criteria:

* Previous adverse reactions to abatacept;
* Known hypersensitivity to abatacept or any of its components;
* Patients at risk of sepsis, such as immunocompromised or HIV positive;
* Patient undergoing a treatment with any other biologic agent;
* Uncontrolled asthma;
* Unstable angina, significant arrhythmia, uncontrolled hypertension, chronic sinusitis, or other chronic or immunological diseases that, in the judgment of the investigator, might interfere with the evaluation, administration of the test drug or pose additional risk to the subject (e.g., gastrointestinal or gastroesophageal disease, chronic infections, scleroderma, hepatic and gallbladder disease, chronic non-allergic pulmonary disease);
* Current users of oral, intramuscular, or intravenous corticosteroids, tricyclic antidepressants or beta-blocker
* Concurrent/prior use of immunomodulatory therapy (within 6 months);
* A diagnosis of eosinophilic esophagitis, eosinophilic colitis, or eosinophilic gastritis;
* Pregnant or breastfeeding women;

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Peanut specific/total IgE at week 24 | 24 weeks
  Relative change in peanut specific/total IgE from baseline to week 24

SECONDARY OUTCOMES:
Peanut-specific IgG4/IgE ratio at week 24 | 24 weeks
  Relative change in peanut-specific IgG4/IgE ratio from baseline to week 24
Peanut-specific IgG4 at week 24 | 24 weeks
  Absolute change in peanut-specific IgG4 from baseline to week 24
Sustained tolerance | Assessed between week 36 and week 48
  Maximum period of avoidance after which a oral food challenge with 300 mg peanut protein is still tolerated
Food dosing reactions | 48 weeks
  Mean cumulative function of food dosing allergic reactions
Desensitization | 36 weeks
  Highest tolerated dose on an oral food challenge at week 36
Desensitization speed | 36 weeks
  Time from the onset of oral immunotherapy to the maintenance dose of 300mg
Adverse events | 48 weeks
  Overall rate of adverse events

OTHER OUTCOMES:
Atopy patch test | week 12, week 24 and week 48
  Change in peanut atopy patch test from baseline
Skin test | week 12, week 24 and week 48
  Change in peanut skin test from baseline
Peanut specific/total IgE, other time points | weeks 2, 6, 12, 36 and 48
  Relative change in peanut specific/total IgE from baseline
Peanut-specific IgG4/IgE ratio, other time points | weeks 2, 6, 12, 36 and 48
  Relative change in peanut-specific IgG4/IgE ratio from baseline
Peanut-specific IgG4, other time points | weeks 2, 6, 12, 36 and 48
  Absolute change from baseline in peanut-specific IgG4

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No